CLINICAL TRIAL: NCT06683482
Title: Ethnographic Study on Advanced Breast Cancer Patients and Their Caregivers in Spain
Brief Title: A Qualitative Study on Advanced Breast Cancer Patients and Their Caregivers in Spain
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-ES-984-6674
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Advanced Breast Cancer Living in Spain and their Caregivers: Participants with different types of breast cancers living in Spain will be observed in this study. Participants will not receive any study drug in this study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No study drug will be administered as a part of this study.

SUMMARY:
The main goal of this ethnographic study is to learn a holistic and enriched view of the behaviors, actions, and views of a group of people with advanced breast cancer (ABC) cancer living in Spain. The primary objective of this study is to collect data on the psychosocial needs of (ABC) patients to identify spaces and strategies to improve these needs.

ELIGIBILITY:
Key Inclusion Criteria:

1. Informed consent to individual in the qualitative study and to allow the recording of the interview for analyses purposes (individual and/or caregiver).
2. Women or men (individual and/or caregiver) over 18 years of age.
3. Confirmed diagnosis of triple-negative breast cancer (TNBC), hormone receptor (HR)+/ human epidermal growth factor receptor 2 (HER2)-, HER2+ unresectable locally advanced breast cancer (ULABC) or metastatic breast cancer (mBC) (individual).
4. Individuals must have initiated at least the firstline treatment.
5. Functional status according to the Eastern Cooperative Oncology Group (ECOG) scale 0-2 (individual).
6. Ability to conduct interviews from home (individual and/or caregiver) or remotely (ie, with technology available for an online interview).

Key Exclusion Criteria:

1. Individual unable to collaborate in the collection of necessary information (alteration in mental status, noncollaboration, limited language comprehension).
2. Individual unable or unwilling to provide informed consent.

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes individuals with BC subtypes in the advanced setting (TNBC, HR+/HER2-, and HER2+ [with any HR]), and also their caregivers will be observed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Responses to the Open-ended questionnaires | Up to 4 weeks
  This qualitative ethnographic study will be carried out through the transcriptions of open-ended interviews. The variables of interest will consist of a set of sociodemographic data, as well as results from emotional and psychological.

SECONDARY OUTCOMES:
Number of Participants with Responses to the Open-ended Questionnaires Related to Intimacy and Sexuality | Up to 4 weeks
Number of Participants With Responses to the Economic Impact of the Disease | Up to 4 weeks
Number of Participants With Responses Open-ended Interviews to Assess Importance of Hereditary BC, Genetic Testing and Generic Counselling in ABC Patients | Up to 4 weeks
Number of Participants With Responses to the Open-ended interviews to assess the Level of Insight and Opportunities for Access to Clinical Studies to Promote Research and Access to Novel Therapeutic Options | Up to 4 weeks
Number of Participants With Responses to the Open-ended Interviews to Assess Whether There is any Difference Between the Analyses of the Above Characteristics by BC Subtype | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- Salvetti & Llombart Sl, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06683482